CLINICAL TRIAL: NCT02331368
Title: Phase 2 Multi-center Study of Anti-Programmed-Death-1 [Anti-PD-1] During Lymphopenic State After High-Dose Chemotherapy and Autologous Hematopoietic Stem Cell Transplant [HDT/ASCT] for Multiple Myeloma
Brief Title: Phase 2 Multi-center Study of Anti-PD-1 During Lymphopenic State After HDT/ASCT for Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2014.134
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Anti-PD-1; Pembrolizumab; Post-transplant; Maintenance
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Lenalidomide; pembrolizumab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti-PD-1 (MK-3475) (Experimental): Standard Treatment:
  High-dose Melphalan and autologous stem cell transplantation with post-transplant maintenance of Lenalidomide.
  Study Treatment:
  200 mg/day of MK-3475 administered every 3 weeks, starting day +14 post-transplant for a total of 9 doses.
  Interventions: Procedure: Autologous Stem Cell Transplant; Drug: Melphalan; Drug: Lenalidomide; Drug: MK-3475

INTERVENTIONS:
Procedure: Autologous Stem Cell Transplant
Drug: Melphalan — 140-200 mg/m^2
Drug: Lenalidomide — 5-15 mg/day starting 45-90 days post-transplant
Drug: MK-3475 — 200 mg/day every 3 weeks starting day +14 post-transplant for a total of 9 doses.
  Other Names: Anti-PD-1; Pembrolizumab

SUMMARY:
Multiple myeloma (MM) is a common incurable blood cancer causing debilitating symptoms-bone pain, kidney failure, low blood counts and infection. Chemotherapy outcomes are disappointing due to short-term response and long-term toxicities.

1. Studies showed these patients have weak immune against MM due to the immune checkpoint mediated by the PD1/PD-L1 interaction between immune cells and MM. Anti-PD-1 antibody (anti-PD1) disrupts this interaction, thus unleashing immune cell function and leading to killing of MM cells.
2. Studies further showed enhancement of this "unleash" after autologous transplant and better MM control by anti-PD1 when used after transplant.
3. Anti-PD1 has been extensively studied in patients with other cancers. It is very safe and effective and has been FDA-approved. Complications are of mild degree and easy to manage successfully in out-patient setting. Severe complications are rare.

Thus, investigators proposed an efficacy study of anti-PD1 treatment after transplant to improve MM treatment outcomes. This was a collaborative study with Medical College of Wisconsin (headquarter of Center for International blood and Marrow Transplant Research). Investigators hypothesized that anti-PD1 treatment would increase the MM response and the MM control duration when added to the standard MM treatment after transplant. Anti-PD1 was given at the dose and interval, which had been studied previously (200 mg intravenous injection every 3 weeks) between 2 weeks until 6 months after transplant. Subjects were monitored closely during and after anti-PD1 therapy until at least 1 year post transplant. Late complications were followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with MM (Multiple Myeloma) of any stage
* Has no Progressive Disease (PD) AND has suboptimal response with primary therapy
* Has measurable disease
* Has no prior hematopoietic stem cell transplant of any type
* Has performance status of 0 or 1 (Eastern Cooperative Oncology, ECOG, Performance Scale)
* Has had a successful peripheral blood stem cell collection with G-CSF (Filgrastim) +/- Plerixafor (Mozobil) only
* Be willing and able to provide written informed consent
* Female subjects of child bearing age should have negative urine or serum pregnancy test
* Female subjects of child bearing age must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity
* Male subjects must agree to use an adequate method of contraception
* Subject must be able to swallow capsules
* Must demonstrate adequate organ function

Exclusion Criteria:

* Has history of repeat infections, amyloidosis, hyperviscosity, plasma cell leukemia, POEMS syndrome, Waldenstrom's macroglobulinemia, non-secretory multiple myeloma, or IgM myeloma
* Has known CNS (Central Nervous System) involvement or history of resolved CNS involvement
* Has an active autoimmune disease or history of autoimmune disease that requires systemic treatment with steroids of immunosuppressive agents.
* Has active, non-infectious pneumonitis
* Has diagnosis of immunosuppressive disorder or on immunosuppressive therapy within 7 days of transplant admission
* Is currently participating in or has previously participated in the study of an investigational drug/device within 4 weeks of transplant admission
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or CTLA-4
* Has had prior monoclonal antibody, chemotherapy, small molecule therapy, or radiation within 2 weeks of transplant admission
* Has not recovered from adverse events due to previously administered agent
* Must be free of additional malignancy for at least 5 years
* Has an active infection requiring systemic therapy
* Has known psychiatric or substance abuse disorders that would interfere with requirements of the study
* Is pregnant or breastfeeding or expecting to conceive
* Has known HIV, Hepatitis B, or Hepatitis C infection
* Has clinically significant coagulopathy
* Has known symptomatic heart failure, unstable angina pectoris, or cardiac arrhythmia
* Has received any type of hematopoietic cell transplant
* Has received a live vaccine within 30 days of transplant admission
* Is or has an immediate family member whos is investigational site or sponsor staff directly involved with this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Attaphol Pawarode, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] D'Souza A, Hari P, Pasquini M, Braun T, Johnson B, Lundy S, Couriel D, Hamadani M, Magenau J, Dhakal B, Shah NN, Riwes M, Parkin B, Reddy P, Pawarode A. A Phase 2 Study of Pembrolizumab during Lymphodepletion after Autologous Hematopoietic Cell Transplantation for Multiple Myeloma. Biol Blood Marrow Transplant. 2019 Aug;25(8):1492-1497. doi: 10.1016/j.bbmt.2019.04.005. Epub 2019 Apr 6. PMID 30959163

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 patients were enrolled and 3 withdrew consent prior to being treated.
Groups:
- Anti-PD-1 (MK-3475): Study Treatment:
  200 mg/day of MK-3475 administered every 3 weeks, starting day +14 post-transplant for a total of 9 doses.
Period: Overall Study
Arm/Group | Anti-PD-1 (MK-3475)
Started | 32
Completed | 29
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: 32 patients were enrolled, however 3 withdrew consent prior to beginning treatment so they were not included in the baseline population analysis.
Arm/Group | Anti-PD-1 (MK-3475)
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 59 [49 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients That Achieve Complete Response
Description: The primary efficacy endpoint is complete response rate. The complete response rate was estimated by the observed proportion of complete responders at day 180. Complete response (CR) was defined as negative immunofixation of serum and urine and disappearance of any soft tissue plasmacytomas, and <5% plasma cells in bone marrow and negative bone marrow flow cytometry.
Time Frame: 180 days post-transplant
Population: 32 patients were enrolled. 3 withdrew consent prior to treatment. Of the 29 treated, 26 were evaluable for response (subjects who received 2-9 doses of MK-3475 were evaluable). Of the 26, 23 completed end-of-treatment response evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-PD-1 (MK-3475)
Number analyzed (Participants) | 23
Participants | 7

2. Secondary Outcome: The Estimated Percentage of Patients Alive Without Relapse or Progression at 2 Years
Description: Progression is defined as an increase of ≥ 25% from the lowest response value in any one or more of the following:
  Serum M-component with an absolute increase ≥ 0.5 g/dL; and/or Urine M-component with an absolute increase ≥ 200 mg/24 hours; and/or Only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels (absolute increase must be >100mg/l) Bone marrow plasma cell percentage (absolute % must be ≥10% Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas Development of hypercalcemia (corrected serum calcium >11.5mg/100ml) that can be attributed solely to the plasma cell proliferative disorder
Time Frame: 2 Years
Population: 32 patients were enrolled. 3 withdrew consent prior to treatment. Of the 29 treated, 26 were evaluable for response (subjects who received 2-9 doses of MK-3475 were evaluable). Of the 26, 23 completed end-of-treatment response evaluation and were included in primary endpoint analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Anti-PD-1 (MK-3475)
Number analyzed (Participants) | 23
percentage of patients | 83 [68 to 100]

3. Secondary Outcome: The Estimated Percentage of Patients Alive at 2 Years
Time Frame: 2 Years
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Anti-PD-1 (MK-3475)
Number analyzed (Participants) | 23
percentage of patients | 100

ADVERSE EVENTS:
Time Frame: All adverse events were recorded from the time the consent form is signed through 30 days following cessation of treatment. Any serious adverse event (SAE), or follow up to a serious adverse event that occurred from the time the consent was signed through 90 days following cessation of treatment, or the initiation of new anti-multiple myeloma therapy (excluding maintenance treatment as specified in this protocol), whichever was earlier, was recorded.
Arm/Group | Anti-PD-1 (MK-3475)
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 14/32
Other Adverse Events (participants affected / at risk) | 30/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-PD-1 (MK-3475) (N=32)
Blood and Lymphatic Disorder, Other (Blood and lymphatic system disorders) | 4 (4)
Infusion related reaction (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Radiculitis (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-PD-1 (MK-3475) (N=32)
Anemia (Blood and lymphatic system disorders) | 18 (75)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 7 (10)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 7 (8)
Hypothyroidism (Endocrine disorders) | 5 (6)
Blurred vision (Eye disorders) | 3 (3)
Cataract (Eye disorders) | 1 (1)
Eye disorders - Other (Eye disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 9 (14)
Diarrhea (Gastrointestinal disorders) | 24 (47)
Dry mouth (Gastrointestinal disorders) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 3 (6)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 19 (26)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (17)
Chills (General disorders) | 2 (3)
Edema limbs (General disorders) | 3 (3)
Fatigue (General disorders) | 19 (28)
Fever (General disorders) | 11 (15)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (3)
Infusion related reaction (General disorders) | 4 (5)
Irritability (General disorders) | 1 (1)
Neck edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Allergic reaction (Immune system disorders) | 1 (1)
Autoimmune disorder (Immune system disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 8 (9)
Urinary tract infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 11 (18)
Alkaline phosphatase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 8 (9)
Blood bilirubin increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 3 (3)
Investigations - Other (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 18 (111)
Lymphocyte count increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 19 (76)
Platelet count decreased (Investigations) | 19 (107)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 3 (3)
White blood cell decreased (Investigations) | 17 (93)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (27)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (4)
Hypernatremia (Metabolism and nutrition disorders) | 2 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 6 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 (27)
Hypocalcemia (Metabolism and nutrition disorders) | 17 (55)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (6)
Hypokalemia (Metabolism and nutrition disorders) | 11 (19)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 8 (21)
Hypophosphatemia (Metabolism and nutrition disorders) | 14 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Dizziness (Nervous system disorders) | 6 (7)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 8 (10)
Memory impairment (Nervous system disorders) | 1 (1)
Movements involuntary (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Radiculitis (Nervous system disorders) | 1 (2)
Sinus pain (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 1 (2)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 5 (5)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (5)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (10)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (10)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 10 (25)
Hypotension (Vascular disorders) | 10 (15)
Thromboembolic event (Vascular disorders) | 2 (3)

LIMITATIONS AND CAVEATS:
The study was terminated during a pending major amendment after interim analysis and until the FDA mandate of the discontinuation of any combination therapy of MK-3475 and lenalidomide.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT02331368/Prot_SAP_000.pdf